CLINICAL TRIAL: NCT00071175
Title: Lupus Genetic Studies; Lupus Family Registry & Repository
Brief Title: Lupus Genetics Studies
Acronym: LFRR
Status: Completed | Type: Observational
Sponsor: Oklahoma Medical Research Foundation (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NIAMS-103; 5P01AR049084-09 (NIH); AI24717; AR42460; AR049084; AR52253; AR62277
Record Dates: First submitted 2003-10-14; First posted 2003-10-15 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Genetics
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA, sera, plasma, cell lines
Oversight: Data Monitoring Committee: No

SUMMARY:
The Lupus Genetics Studies and Lupus Family Registry & Repository are working to find the genes that reveal the causes of systemic lupus erythematosus (SLE, or lupus). The study is enrolling families of all ethnic backgrounds from the United States, Canada, Puerto Rico, and the Virgin Islands that have one or more living members diagnosed with SLE.

DETAILED DESCRIPTION:
SLE is an often crippling and potentially fatal autoimmune disease that is nine times more prevalent in women than in men, and four times more likely to affect African American females than Caucasian females. It is suspected that a genetic predisposition along with environmental factors contribute to the clinical manifestation of SLE. The Lupus Genetics Studies consist of several familial SLE studies, including the Lupus Family Registry & Repository (LFRR, formerly known as the Lupus Multiplex Registry & Repository, or LMRR). The Lupus Studies enroll families of all ethnicities with one or more members diagnosed with systemic lupus to determine what genes contribute to the development of the disease.

Additionally, the Lupus Family Registry & Repository is the largest repository of its kind in North America. In addition to the research done on site, the Repository serves as a national resource for scientists interested in conducting research on SLE and families either simplex or multiplex for lupus. Data, serum samples, and DNA samples are available to researchers. By collecting families in which two or more living individuals have been diagnosed with SLE, the study is utilizing the genetic link between the affected family members to discover disease-associated genes.

Records will be requested from the patients' treating physicians to document various lupus symptoms and related problems. One-time blood samples will be collected from the patients as well as from certain family members and an unrelated volunteer. There is no cost to participate and the study pays for sample draws and shipping.

ELIGIBILITY:
Inclusion Criteria:

* Families in which one or more living members have been diagnosed with systemic lupus erythematosus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with SLE Families with living members diagnosed with SLE
Sampling Method: Non-Probability Sample
Enrollment: 3460 (Actual)
Dates: Start 1995-10; Primary Completion 2012-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B. Harley, MD, PhD, Principal Investigator — Member & Program Head, Arthritis and Immunology Research Program; Oklahoma Medical Research Foundation
Locations (1):
- Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Lee YH, Rho YH, Choi SJ, Ji JD, Song GG, Nath SK, Harley JB. The PTPN22 C1858T functional polymorphism and autoimmune diseases--a meta-analysis. Rheumatology (Oxford). 2007 Jan;46(1):49-56. doi: 10.1093/rheumatology/kel170. Epub 2006 Jun 7. PMID 16760194
- [Background] Xing C, Sestak AL, Kelly JA, Nguyen KL, Bruner GR, Harley JB, Gray-McGuire C. Localization and replication of the systemic lupus erythematosus linkage signal at 4p16: interaction with 2p11, 12q24 and 19q13 in European Americans. Hum Genet. 2007 Jan;120(5):623-31. doi: 10.1007/s00439-006-0248-4. Epub 2006 Sep 16. PMID 16983533
- [Background] Harley JB, Kelly JA, Kaufman KM. Unraveling the genetics of systemic lupus erythematosus. Springer Semin Immunopathol. 2006 Oct;28(2):119-30. doi: 10.1007/s00281-006-0040-5. Epub 2006 Sep 22. PMID 17021721
- [Background] Forabosco P, Gorman JD, Cleveland C, Kelly JA, Fisher SA, Ortmann WA, Johansson C, Johanneson B, Moser KL, Gaffney PM, Tsao BP, Cantor RM, Alarcon-Riquelme ME, Behrens TW, Harley JB, Lewis CM, Criswell LA. Meta-analysis of genome-wide linkage studies of systemic lupus erythematosus. Genes Immun. 2006 Oct;7(7):609-14. doi: 10.1038/sj.gene.6364338. Epub 2006 Sep 14. PMID 16971955
- [Background] Scofield RH, Bruner GR, Harley JB, Namjou B. Autoimmune thyroid disease is associated with a diagnosis of secondary Sjogren's syndrome in familial systemic lupus. Ann Rheum Dis. 2007 Mar;66(3):410-3. doi: 10.1136/ard.2006.055103. Epub 2006 Sep 19. PMID 16984944
- [Background] Kaufman KM, Kelly JA, Herring BJ, Adler AJ, Glenn SB, Namjou B, Frank SG, Dawson SL, Bruner GR, James JA, Harley JB. Evaluation of the genetic association of the PTPN22 R620W polymorphism in familial and sporadic systemic lupus erythematosus. Arthritis Rheum. 2006 Aug;54(8):2533-40. doi: 10.1002/art.21963. PMID 16868974
- [Background] Ramos PS, Kelly JA, Gray-McGuire C, Bruner GR, Leiran AN, Meyer CM, Namjou B, Espe KJ, Ortmann WA, Reichlin M, Langefeld CD, James JA, Gaffney PM, Behrens TW, Harley JB, Moser KL. Familial aggregation and linkage analysis of autoantibody traits in pedigrees multiplex for systemic lupus erythematosus. Genes Immun. 2006 Jul;7(5):417-32. doi: 10.1038/sj.gene.6364316. Epub 2006 Jun 15. PMID 16775618
- [Background] Lee YH, Harley JB, Nath SK. Meta-analysis of TNF-alpha promoter -308 A/G polymorphism and SLE susceptibility. Eur J Hum Genet. 2006 Mar;14(3):364-71. doi: 10.1038/sj.ejhg.5201566. PMID 16418737
- [Background] Nolsoe RL, Kelly JA, Pociot F, Moser KL, Kristiansen OP, Mandrup-Poulsen T, Harley JB. Functional promoter haplotypes of the human FAS gene are associated with the phenotype of SLE characterized by thrombocytopenia. Genes Immun. 2005 Dec;6(8):699-706. doi: 10.1038/sj.gene.6364259. PMID 16163374
- [Background] Xing C, Gray-McGuire C, Kelly JA, Garriott P, Bukulmez H, Harley JB, Olson JM. Genetic linkage of systemic lupus erythematosus to 13q32 in African American families with affected male members. Hum Genet. 2005 Dec;118(3-4):309-21. doi: 10.1007/s00439-005-0061-5. Epub 2005 Sep 28. PMID 16189706
- [Background] Lee YH, Witte T, Momot T, Schmidt RE, Kaufman KM, Harley JB, Sestak AL. The mannose-binding lectin gene polymorphisms and systemic lupus erythematosus: two case-control studies and a meta-analysis. Arthritis Rheum. 2005 Dec;52(12):3966-74. doi: 10.1002/art.21484. PMID 16320344
- [Background] Namjou B, Kelly JA, Kilpatrick J, Kaufman KM, Nath SK, Scofield RH, Harley JB. Linkage at 5q14.3-15 in multiplex systemic lupus erythematosus pedigrees stratified by autoimmune thyroid disease. Arthritis Rheum. 2005 Nov;52(11):3646-50. doi: 10.1002/art.21413. PMID 16255059
- [Background] Sestak AL, Nath SK, Harley JB. Genetics of systemic lupus erythematosus: how far have we come? Rheum Dis Clin North Am. 2005 May;31(2):223-44, v. doi: 10.1016/j.rdc.2005.01.005. PMID 15922143
- [Result] Harley JB, Moser KL, Gaffney PM, Behrens TW. The genetics of human systemic lupus erythematosus. Curr Opin Immunol. 1998 Dec;10(6):690-6. doi: 10.1016/s0952-7915(98)80090-3. PMID 9914226
- [Result] Moser KL, Gray-McGuire C, Kelly J, Asundi N, Yu H, Bruner GR, Mange M, Hogue R, Neas BR, Harley JB. Confirmation of genetic linkage between human systemic lupus erythematosus and chromosome 1q41. Arthritis Rheum. 1999 Sep;42(9):1902-7. doi: 10.1002/1529-0131(199909)42:93.0.CO;2-G. PMID 10513806
- [Result] Rao S, Olson JM, Moser KL, Gray-McGuire C, Bruner GR, Kelly J, Harley JB. Linkage analysis of human systemic lupus erythematosus-related traits: a principal component approach. Arthritis Rheum. 2001 Dec;44(12):2807-18. doi: 10.1002/1529-0131(200112)44:123.0.co;2-c. PMID 11762941
- [Result] Tsao BP, Grossman JM, Riemekasten G, Strong N, Kalsi J, Wallace DJ, Chen CJ, Lau CS, Ginzler EM, Goldstein R, Kalunian KC, Harley JB, Arnett FC, Hahn BH, Cantor RM. Familiality and co-occurrence of clinical features of systemic lupus erythematosus. Arthritis Rheum. 2002 Oct;46(10):2678-85. doi: 10.1002/art.10519. PMID 12384927
- [Result] Namjou B, Nath SK, Kilpatrick J, Kelly JA, Reid J, James JA, Harley JB. Stratification of pedigrees multiplex for systemic lupus erythematosus and for self-reported rheumatoid arthritis detects a systemic lupus erythematosus susceptibility gene (SLER1) at 5p15.3. Arthritis Rheum. 2002 Nov;46(11):2937-45. doi: 10.1002/art.10588. PMID 12428235
- [Result] Scofield RH, Bruner GR, Kelly JA, Kilpatrick J, Bacino D, Nath SK, Harley JB. Thrombocytopenia identifies a severe familial phenotype of systemic lupus erythematosus and reveals genetic linkages at 1q22 and 11p13. Blood. 2003 Feb 1;101(3):992-7. doi: 10.1182/blood-2002-04-1003. Epub 2002 Sep 12. PMID 12393658
- [Result] Heinlen LD, McClain MT, Kim X, Quintero DR, James JA, Harley JB, Scofield RH. Anti-Ro and anti-nRNP response in unaffected family members of SLE patients. Lupus. 2003;12(4):335-7. doi: 10.1191/0961203303lu377xx. No abstract available. PMID 12729062
- [Result] Nath SK, Quintero-Del-Rio AI, Kilpatrick J, Feo L, Ballesteros M, Harley JB. Linkage at 12q24 with systemic lupus erythematosus (SLE) is established and confirmed in Hispanic and European American families. Am J Hum Genet. 2004 Jan;74(1):73-82. doi: 10.1086/380913. Epub 2003 Dec 4. PMID 14658095
- [Result] Nath SK, Kilpatrick J, Harley JB. Genetics of human systemic lupus erythematosus: the emerging picture. Curr Opin Immunol. 2004 Dec;16(6):794-800. doi: 10.1016/j.coi.2004.09.007. PMID 15511675
- [Result] Sawalha AH, Harley JB. Antinuclear autoantibodies in systemic lupus erythematosus. Curr Opin Rheumatol. 2004 Sep;16(5):534-40. doi: 10.1097/01.bor.0000135452.62800.8f. PMID 15314490
- [Result] Quintero-del-Rio AI, Kelly JA, Garriott CP, Hutchings DC, Frank SG, Aston CE, Harley JB. SLEN2 (2q34-35) and SLEN1 (10q22.3) replication in systemic lupus erythematosus stratified by nephritis. Am J Hum Genet. 2004 Aug;75(2):346-8. doi: 10.1086/422460. No abstract available. PMID 15307049
- [Result] Sawalha AH, Schmid WR, Binder SR, Bacino DK, Harley JB. Association between systemic lupus erythematosus and Helicobacter pylori seronegativity. J Rheumatol. 2004 Aug;31(8):1546-50. PMID 15290733
- [Result] Nath SK, Kelly JA, Harley JB, Scofield RH. Mapping the systematic lupus erythematosus susceptibility genes. Methods Mol Med. 2004;102:11-29. doi: 10.1385/1-59259-805-6:011. PMID 15286378
- [Result] Nath SK, Namjou B, Garriott CP, Frank S, Joslin PA, Kilpatrick J, Kelly JA, Harley JB. Linkage analysis of SLE susceptibility: confirmation of SLER1 at 5p15.3. Genes Immun. 2004 May;5(3):209-14. doi: 10.1038/sj.gene.6364060. PMID 15014430
- [Result] Nath SK, Namjou B, Kilpatrick J, Garriott CP, Bruner GR, Scofield RH, Harley JB. A candidate region on 11p13 for systemic lupus erythematosus: a linkage identified in African-American families. J Investig Dermatol Symp Proc. 2004 Jan;9(1):64-7. doi: 10.1111/j.1087-0024.2004.00830.x. PMID 14870988
- [Result] Nath SK, Namjou B, Hutchings D, Garriott CP, Pongratz C, Guthridge J, James JA. Systemic lupus erythematosus (SLE) and chromosome 16: confirmation of linkage to 16q12-13 and evidence for genetic heterogeneity. Eur J Hum Genet. 2004 Aug;12(8):668-72. doi: 10.1038/sj.ejhg.5201209. PMID 15114372
- [Result] Lee YH, Harley JB, Nath SK. CTLA-4 polymorphisms and systemic lupus erythematosus (SLE): a meta-analysis. Hum Genet. 2005 Apr;116(5):361-7. doi: 10.1007/s00439-004-1244-1. Epub 2005 Feb 2. PMID 15688186
- [Result] Kochi Y, Yamada R, Suzuki A, Harley JB, Shirasawa S, Sawada T, Bae SC, Tokuhiro S, Chang X, Sekine A, Takahashi A, Tsunoda T, Ohnishi Y, Kaufman KM, Kang CP, Kang C, Otsubo S, Yumura W, Mimori A, Koike T, Nakamura Y, Sasazuki T, Yamamoto K. A functional variant in FCRL3, encoding Fc receptor-like 3, is associated with rheumatoid arthritis and several autoimmunities. Nat Genet. 2005 May;37(5):478-85. doi: 10.1038/ng1540. Epub 2005 Apr 17. PMID 15838509
- See also: Lupus Family Registry & Repository Webpage: For potential participants and researchers — http://lupus.omrf.org